CLINICAL TRIAL: NCT04354922
Title: Effects of Different Exercising Intensities and Frequencies of Walking Exercise on Depressive Mood and Insomnia in Older Adults
Brief Title: Different Exercising Intensities and Frequencies of Exercise on Depressive Mood and Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DI
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-07

CONDITIONS: Sleep Disorder; Depressive Symptoms
Keywords: Insomnia; Mood; Exercise
MeSH Terms: conditions — Sleep Wake Disorders; Depression; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: 5 groups ×2 times factorial design
Who Masked: Outcomes Assessor
Masking Description: Single-blind (Outcome Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Attention control (Placebo Comparator): Subjects in this group will receive one session of 75 minutes stretching exercise per week throughout the 12 weeks experimental period
  Interventions: Behavioral: Exercise intervention
- Moderate-intensity walking exercise ×3/wk (Active Comparator): Subjects in this group will receive three sessions of 50 minutes vigorous walking exercise per week throughout the 12 weeks experimental period
  Interventions: Behavioral: Exercise intervention
- Moderate-intensity walking exercise ×1/wk (Active Comparator): Subjects in this group will receive one session of 150 minutes vigorous walking exercise per week throughout the 12 weeks experimental period
  Interventions: Behavioral: Exercise intervention
- Vigorous-intensity walking exercise ×3/wk (Active Comparator): Subjects in this group will receive three sessions of 25 minutes vigorous walking exercise per week throughout the 12 weeks experimental period
  Interventions: Behavioral: Exercise intervention
- Vigorous-intensity walking exercise ×1/wk (Active Comparator): Subjects in this group will receive one session of 75 minutes vigorous walking exercise per week throughout the 12 weeks experimental period
  Interventions: Behavioral: Exercise intervention

INTERVENTIONS:
Behavioral: Exercise intervention — Subjects in attention control group will receive one session of 75 minutes of stretching exercise weekly. All walking exercise session will be performed on motor-driven treadmill. Subjects in moderate-intensity walking groups will walk at an intensity of 3.25 metabolic equivalents (METs). Subjects in vigorous-intensity walking groups will brisk walk at an intensity of 6.5 metabolic equivalents (METs). Warm-up and cool-down will be provided before and after the training. Participants who failed to achieve 80% attendance will be excluded from the study. All exercise sessions were supervised by qualified athletic coach.

SUMMARY:
Aerobic exercise intervention for depression was conventionally recommended three times weekly with moderate intensity in previous studies, but little is known about the training effect of aerobic exercise at low frequency and vigorous intensity. The purpose of this study is to compare the training effect of aerobic exercise at different exercising frequencies and intensities on older adults with comorbid insomnia and depressive symptoms. In this study, the investigators will investigate two types of aerobic exercise (i.e., vigorous-intensity exercise and moderate-intensity exercise) under different exercising frequencies (i.e., regular exercising pattern and weekend warrior). Individuals with chronic insomnia and depressive symptoms will be recruited and randomly allocated into 5 groups: 1) attention control group (stretching exercise), 2) moderate intensity exercise performed thrice weekly (MIE×3/wk), 3) moderate intensity exercise performed once weekly (MIE×1/wk), 4) vigorous intensity exercise performed thrice weekly (VIE×3/wk), and 5) vigorous intensity exercise performed once weekly (VIE×1/wk). Intervention will be maintained for 12 weeks. Outcome assessments will be conducted at baseline, 6 weeks and 12 weeks after the intervention. Outcomes including depressive status, chronic insomnia, objective sleep quality and pattern (measured by Actigraphy), subjective sleep quality (measured by Epworth sleepiness scale, insomnia severity index, PSQI), anxiety status (measured by HADS and GAD-7), quality of life (measured by SF-12), attention level (measured by computer attention test), exercise enjoyment (measured by physical activity enjoyment scale), habitual physical activity level (measured by IPAQ), aerobic fitness (measured by metabolic cart), body adiposity (measured by DXA), blood chemistry, adherence, medication usage, and adverse events will be measure in this study. This proposed study will provide pilot evidence for the benefits, effectiveness, safety, adherence, and sustainability of low-frequency vigorous aerobic exercise. the investigators expect the low-frequency exercise modality will enhance the practical suitability of aerobic exercise and will provide evidence for weekend warrior aerobic training strategy as a new exercise option in the management of elderly insomnia and depression.

ELIGIBILITY:
Inclusion Criteria:

1. borderline abnormal depression with score above 8 out of 21 on Hospital Anxiety and Depression Scale (HADS),
2. chronic insomnia according to the fifth edition of the diagnostic and statistical manual of mental disorder (DSM-5),
3. Cantonese, Mandarin or English speaking, and 4) age 50 or above. To enhance generalizability, males and females will be recruited.

Exclusion Criteria:

1. contraindications to participating in physical exercise;
2. regular exercise habit in the past three months (i.e.,>75 minutes of vigorous-intensity exercise weekly or >150 minutes of moderate-intensity exercise weekly);
3. any pre-existing medical or physical issues that affect the experimental test and exercise intervention;
4. diagnosis with psychosis, schizophrenia or bipolar disorder;
5. currently receiving non-medication treatment for depression or insomnia, such as mindfulness training or cognitive behavior therapy;
6. shift worker or other commitment that interferes with the regular sleep pattern at night; and
7. abnormal heart's electrical activity according to the exercise electrocardiography (ECG) test, such as irregular heartbeat, arrhythmia, and myocardial infarction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Level of depression | After completion of the 12 weeks intervention
  Hospital Anxiety and Depression Scale (HADS) will be used to measure the level of depression
Remission rate of insomnia | After completion of the 12 weeks intervention
  Brief insomnia questionnaire (BIQ) will be employed to diagnose the chronic insomnia based on the DSM-5 criteria.

SECONDARY OUTCOMES:
Subjective sleep data | After completion of the 12 weeks intervention
  The Epworth sleepiness scale, insomnia severity index, and Pittsburgh sleep quality index (PSQI) will be used to measure the sleep quality.
Objective sleep data | After completion of the 12 weeks intervention
  Actigraphy will be used to measure the sleep quality and pattern.
Change in dose of Sleep Medication | After completion of the 12 weeks intervention
  The dose of sleep medication used by the subjects changes after intervention.
7-day Sleep Diary | After completion of the 12 weeks intervention
  Self-recorded sleep parameters (sleep onset latency, sleep efficiency, total sleep time, wake time after sleep onset, number of awakening and average awaken time)
Treatment response rate | After completion of the 12 weeks intervention
  The percentage of participants that have their Score of Pittsburgh Sleep Quality Index reduced by at least 5 points
Body composition | After completion of the 12 weeks intervention
  Body lean mass, fat mass, and bone density will be measured by dual-energy X-ray absorptiometry
Maximal oxygen consumption | After completion of the 12 weeks intervention
  Metabolic cart will measure the maximal oxygen consumption during the maximal exercise test
Anxiety level | After completion of the 12 weeks intervention
  Anxiety level will be measured by HASD and General Anxiety Disorder-7.
Severity of depression | After completion of the 12 weeks intervention
  PHQ-9 will be used to examine the severity of depression.
Blood chemistry tests | After completion of the 12 weeks intervention
  biological markers related to depression and sleep will be measured by enzyme-linked immunosorbent assa
Subjectively measured quality of life | After completion of the 12 weeks intervention
  Measured by the 12-item Short Form Survey, scores range from 0 to 100, higher scores indicating better physical and mental health functioning
Enjoyment of exercise intervention | After completion of the 12 weeks intervention
  Physical activity enjoyment scale will be used to test the subject's perception of the exercise, higher scores reflect greater levels of enjoyment
Attention level | After completion of the 12 weeks intervention
  Computer attention test in PsychoPy v2 software will be employed to measure the attention.
Habitual physical activity | After completion of the 12 weeks intervention
  Habitual physical activity will be measured by IPAQ

CONTACTS AND LOCATIONS:
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chin EC, Yu AP, Leung CK, Bernal JD, Au WW, Fong DY, Cheng CP, Siu PM. Effects of Exercise Frequency and Intensity on Reducing Depressive Symptoms in Older Adults With Insomnia: A Pilot Randomized Controlled Trial. Front Physiol. 2022 Apr 5;13:863457. doi: 10.3389/fphys.2022.863457. eCollection 2022. PMID 35450161